CLINICAL TRIAL: NCT03932864
Title: A Randomized, Placebo-Controlled, Ascending Dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Parameters of MGTA-145 in Healthy Subjects Administered as a Single Agent, as Well as in Combination With Plerixafor
Brief Title: Study Assessing Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MGTA-145 in Healthy Volunteers as a Single Agent or in Combination With Plerixafor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensoma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 145-HV-101
Record Dates: First submitted 2019-04-22; First posted 2019-05-01 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose of MGTA-145 or placebo (Placebo Comparator): MGTA-145 or placebo dose escalation as single agent, single dose
  Interventions: Biological: MGTA-145; Biological: Placebo
- Single Dose MGTA-145 or placebo plus plerixafor (Placebo Comparator): MGTA-145 or placebo in combination with plerixafor, single dose
  Interventions: Biological: MGTA-145; Biological: plerixafor; Biological: Placebo
- Single dose MGTA-145 plus plerixafor for 2 sequential d (Experimental): MGTA-145 in combination with plerixafor on two consecutive days; single dose per day
  Interventions: Biological: MGTA-145; Biological: plerixafor
- Single dose MGTA-145 plus plerixafor followed by apheresis (Experimental): MGTA-145 in combination with plerixafor followed by apheresis
  Interventions: Biological: MGTA-145; Biological: plerixafor

INTERVENTIONS:
Biological: MGTA-145 — MGTA-145 will be given in various doses intravenously
Biological: plerixafor — 240 µg/kg subcutaneously
  Other Names: Mozobil
  Arms: Single Dose MGTA-145 or placebo plus plerixafor; Single dose MGTA-145 plus plerixafor followed by apheresis; Single dose MGTA-145 plus plerixafor for 2 sequential d
Biological: Placebo — Placebo will be given in various doses intravenously
  Arms: Single Ascending Dose of MGTA-145 or placebo; Single Dose MGTA-145 or placebo plus plerixafor

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MGTA-145 in healthy volunteers as a single agent and in combination with plerixafor.

DETAILED DESCRIPTION:
The study consists of up to four parts: Part A, to investigate the safety and tolerability of MGTA-145; Part B, to investigate the safety and tolerability of MGTA-145 when administered in combination with plerixafor; Part C, to investigate the safety and tolerability of two sequential days of dosing MGTA-145 in combination with plerixafor; and Part D, to investigate the safety, tolerability, and measure by apheresis, the total number of CD34+ cells mobilized after a dose of MGTA-145 administered in combination with plerixafor.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 60 years
2. Body weight ≥50 kg and body mass index 19 to 33 kg/m2
3. No clinically significant abnormalities on physical examination at Screening
4. Non-smoker for at least 2 years
5. No clinically significant lab abnormalities for renal, hepatic or hematologic parameters
6. No clinically significant abnormalities on ECG
7. Female subjects must be of non-childbearing potential
8. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception
9. No contraindications for apheresis

Exclusion Criteria:

1. Any clinically significant laboratory value outside the normal range at screening
2. Donation of more than 500 mL of blood or plasma within 12 weeks prior to dosing
3. History of alcoholism or drug abuse within the past 3 years
4. Subject has used any prescription drugs within 14 days prior to dosing or any dietary supplements or non-prescription drugs within 7 days prior to dosing
5. Acute illness, infection (requiring medical treatment [eg, antibiotics]), or surgery within 4 weeks of dosing
6. Seropositive for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus
7. Subject has received another investigational drug or participated in an investigational drug or device study within 12 weeks prior to dosing
8. History of anaphylaxis or clinically important reaction to any drug including plerixafor
9. Any clinically significant hematologic, cardiovascular, pulmonary, central nervous system, metabolic, renal, hepatic, or gastrointestinal conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Safety as measured by incidence of treatment-emergent adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs). | 28 days
  Investigate the safety and tolerability of MGTA-145 following intravenous (IV) administration as monotherapy or in combination with plerixafor in healthy subjects (e.g. adverse events, clinical laboratory tests, vital signs, ECGs)

SECONDARY OUTCOMES:
Pharmacokinetics Biomarkers | 15 days
  Investigate area under the curve (AUC) of MGTA-145
Pharmacokinetics Biomarkers | 15 days
  Investigate maximum plasma concentration (Cmax) of MGTA-145
Pharmacokinetic Biomarkers | 15 days
  Investigate clearance (CL) of MGTA-145
Pharmacokinetic Biomarkers | 15 days
  Investigate the volume of distribution at steady state (Vdss) of MGTA-145
Pharmacokinetic Biomarkers | 15 days
  Investigate the half-life of MGTA-145
Pharmacodynamic Biomarkers | 15 days
  Assess CD34+ cells per uL of blood by flow cytometry
Pharmacodynamic Biomarkers | 15 days
  Assess stem cell progenitors (colony forming units)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace CPU, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No